CLINICAL TRIAL: NCT02595112
Title: Study of Staphylococcus Aureus Colonization of the Posterior Nasal Cavity in Patients Undergoing Otorhinolaryngologic Surgery. A Monocentric Study
Brief Title: Study of Staphylococcus Aureus Colonization of the Posterior Nasal Cavity in Patients Undergoing Otorhinolaryngologic Surgery
Acronym: SREENSTAPH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1508154; 2015-A01620-49 (Other: ANSM)
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2017-12

CONDITIONS: Staphylococcal Infections
Keywords: staphylococcal infections; nasal carriage; nasal cavity; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient undergoing otorhinolaryngologic surgery (Experimental): Staphylococcus aureus carriage is measured in the vestibulum nasi and posterior nasal cavity. Posterior nasal cavity is measured during endoscopic procedure.
  Interventions: Other: Staphylococcus aureus carriage

INTERVENTIONS:
Other: Staphylococcus aureus carriage — Vestibulum nasi and posterior nasal cavity sampling with swabs and posterior nasal cavity sampling by endoscopic procedure during otorhinolaryngologic surgery

SUMMARY:
Staphylococcus aureus nasal carriage is a major risk factor of infection with this bacterium. Staphylococcus aureus colonization of the posterior nasal cavity is still misunderstood. This study is aimed at evaluating the relationship between Staphylococcus aureus strains colonizing the vestibulum nasi, the sphenoethmoidal recess and the nasopharynx.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing otorhinolaryngologic surgery, unknown Staphylococcus aureus carriage state
* Patient affiliated to French Social Security
* Written consent

Exclusion Criteria:

* Antibiotherapy or infectious episode during the month prior enrollment
* coagulation disorder
* neoplasia of the nasal cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
number of patients with staphylococcus aureus carriage in the posterior nasal cavity | Day 1

SECONDARY OUTCOMES:
number of patients with staphylococcus aureus carriage in the vestibulum nasi | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Paul Verhoeven, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No